CLINICAL TRIAL: NCT07040228
Title: A Phase Ib/II Clinical Study of Regorafenib Combined With Toripalimab and Albumin-bound Paclitaxel for the Third-line Treatment of Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Collaborators: Qilu Pharmaceutical Group Co., Ltd (Unknown); Shanghai Junshi Biomedical Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YW2025-28-1
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: Efficacy; Safety; Advanced pancreatic cancer; Regorafenib; Toripalimab
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Scheme Experimental Group (Experimental): Three line treatment of advanced pancreatic cancer with regofinil combined with teripril monoclonal antibody and albumin paclitaxel
  Interventions: Drug: Regorafenib combined with Toripalimab and Albumin paclitaxel

INTERVENTIONS:
Drug: Regorafenib combined with Toripalimab and Albumin paclitaxel — Regorafenib combined with Toripalimab and Albumin paclitaxel as the third line treatment for patients with advanced pancreatic cancer

SUMMARY:
The purpose of this clinical trial is to explore the efficacy and safety of Regorafenib combined with Toripalimab and Paclitaxel-albumin in patients as the third line treatment for patients with unresectable or metastatic pancreatic cancer.The main question it aims to answer is:

Phase Ib: Evaluate the maximum tolerated dose (MTD) of regorafenib and/or phase II clinical recommendations Dose (RP2D).

Phase II: Evaluation of the efficacy and safety of Regorafenib Combined with Terriptylimab and Albumin Paclitaxel for Late Third Line Treatment for pancreatic cancer patients.

Participants will:

Phase Ib: Selected patients will receive treatment with Regorafenib at main dose levels of 40, 80, and 120mg/d (po d1-14 Q3W), Toripalimab(240mg, ivgtt, d1, Q3W), and Paclitaxel-albumi(125mg/m2, ivgtt, d1, 8, Q3W) until disease progression or intolerable toxicity occurs.

Phase II: Regorafenib: Based on the results of the completed Phase I study, determine the dosage for Phase II (po d1-14 Q3W). Toripalimab (240mg, ivgtt, d1, Q3W) and Paclitaxel-albumi (125mg/m2, ivgtt, d1, 8, Q3W) until disease progression or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. The patient fully understands this study, voluntarily participates and signs an informed consent form (ICF);
2. Age ≥ 18 years old and ≤ 80 years old;
3. Patients with unresectable/metastatic pancreatic cancer confirmed by histopathology;
4. Imaging confirmation of tumor progression after previous first-line and second-line standard treatment;
5. According to RECIST 1.1 criteria, patients must have at least one measurable target lesion;
6. Eastern Cancer Collaboration Group (ECOG) Physical Fitness Status Score: 0-2 points;
7. Expected survival time ≥ 2 months;
8. Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9/L, platelets ≥ 100 × 10 ^ 9/L, and hemoglobin ≥ 90 g/L (No blood transfusion or blood products within 14 days prior to laboratory examination.

   Not treated with granulocyte colony-stimulating factor or other hematopoietic stimulating factors);
9. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and ALT ≤ 2.5 times the upper limit of normal values (≤ 5 times the upper limit of normal values for patients with liver metastases); Total bilirubin ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver metastasis);
10. Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result must be negative, And willing to use appropriate contraception methods during the trial period and 6 months after the last administration of the trial drug.

Exclusion Criteria:

1. Have hypersensitivity reactions to any research drug or its components;
2. Concurrent serious uncontrolled infections or other serious uncontrolled accompanying diseases, moderate or severe kidney injury; (such as progressive infection, uncontrollable hypertension, diabetes, etc.);
3. Heart function and disease meet one of the following conditions:

   1. Long QTc syndrome or QTc interval>480 ms;
   2. Complete left bundle branch block, grade II or III atrioventricular block;
   3. Severe and uncontrolled arrhythmias requiring medication treatment;
   4. New York College of Cardiology classification ≥ III;
   5. Heart ejection fraction (LVEF) below 50%;
   6. History of myocardial infarction, unstable angina, and severe unstable ventricular arrhythmia within 6 months prior to recruitment or any other arrhythmia requiring treatment, history of clinically severe pericardial disease, or there may be electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
4. Active infection of hepatitis B and C (hepatitis B virus surface antigen is positive and hepatitis B virus DNA exceeds 1x103 copies/mL; Hepatitis C virus RNA exceeding 1x103 copies/mL).Asymptomatic chronic carriers of hepatitis B or hepatitis C excluded;
5. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
6. Imaging confirms intestinal obstruction;
7. Previously or currently suffering from other malignant tumors simultaneously (Except for non melanoma basal cell carcinoma and breast/cervical carcinoma in situ that have been effectively controlled and other malignant tumors that have been effectively controlled without treatment in the past five years);
8. Pregnant and lactating women, as well as reproductive age patients who are unwilling to take contraceptive measures;
9. Patients who require treatment for merging with other malignant tumors;
10. History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as at least 2.5mL of bright red blood) within one month prior to the first administration;
11. Within 6 months prior to the first administration, there are arterial embolism, severe bleeding (excluding bleeding caused by surgery), and a tendency for severe bleeding;
12. Merge symptomatic brain metastases, meningeal metastases, spinal cord tumor invasion, and spinal cord compression syndrome;
13. Have used other clinical trial drugs within one month before the first administration;
14. The researchers have determined that patients who are not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
(PFS) | Dated from the first treatment with study medication to the first documented PD or death owing to any cause, whichever occurred first,assessed up to 60 months.
  Progression-Free Survival

SECONDARY OUTCOMES:
ORR | up to 60 months
  Objective Response Rate
OS | Dated from the date of first treatment with study medication to the date of death owing to any cause or censored on the date of last follow-up,assessed up to 60 months.
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided